CLINICAL TRIAL: NCT02395484
Title: Species and Metagenome Analysis of Gut Microbiota in Chronic Constipation Patients
Brief Title: Metagenome Analysis of Gut Microbiota in CC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, MD, Jinling Hospital, China
Other Study IDs: MetagenomeNanjing
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- constipation: collect stool samples from constipation patients
- healthy controls: collect stool samples from healthy controls patients

SUMMARY:
Constipation is a heterogeneous and multifactorial disease, influenced by a number of different genetic and environmental factors. By applying the standard two-stage GWAS strategy to design and carry out a metagenome-wide association study (MGWAS) to find the relationship between gut microbiota and constipation, to identify disease-associated metagenomic markers.

DETAILED DESCRIPTION:
This study is a two-stage case-control metagenome-wide association study (MGWAS) based on deep next-generation shotgun sequencing of DNA extracted from the stool samples from a total of 50 Chinese constipation patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic constipation according to Rome III criteria;
2. Age ≥ 18 years;
3. BMI: 18.5-25kg/m2;

Exclusion Criteria:

1. Bowel constipation due to innate factor (e.g. megacolon) or secondary interventions (e.g. drugs, endocrine, metabolic, neurologic or psychologic disorders);
2. History or evidence of gastrointestinal diseases (e.g. cancer, inflammatory bowel diseases);
3. Previous abdominal surgery, except cholecystectomy, appendicectomy, tubal ligation and cesarean section;
4. Previous proctological or perianal surgery;
5. Rectal prolapse and/or grade 3-4 internal hemorrhoids according to AGA classification;
6. A constipation condition meeting the Rome III criteria for IBS or functional abdominal pain syndrome;
7. Pregnant or breast-feeding women;
8. Infection with enteric pathogen;
9. Usage of probiotics, prebiotics, antibiotics or PPIs within the last month;
10. Smoking or alcohol addiction within the last 3 months;
11. Uncontrolled hepatic, renal, cardiovascular, respiratory or psychiatric disease;
12. Disease or therapy with drugs (e.g. antidepressants, opioid narcotic analgesics, anticholinergics, calcium antagonists, nitrates, antimuscarinics) that, in the opinion of the investigator, could affect intestinal transit and microbiota.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 faecal samples were obtained from constipation patients and 50 faecal samples were obtained from healthy volunteers
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
taxonomic and functional characterization of gut microbiota | one year

SECONDARY OUTCOMES:
Gut-microbiota-based constipation classification | one year
constipation-associated gut microbial markers | one year

CONTACTS AND LOCATIONS:
Overall Officials: Chao Ding, MD, Principal Investigator — Department of Generay Surgery, Jinling hospital; Hongliang Tian, PhD, Principal Investigator — Department of Generay Surgery, Jinling hospital
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China